CLINICAL TRIAL: NCT00259363
Title: Phase I-II Study of Preoperative Oxaliplatin-FU and Radiotherapy for Patients With Rectal Cancer
Brief Title: Oxaliplatin in Rectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study cancelled because recruitment rate was too slow
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8330
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin — oxaliplatin 60/mg/m2/15 days, 5-FU 225 mg/m2/day 5 weeks during radiotherapy (RT) 45 Gys/25 days

SUMMARY:
* Phase I: To determine the maximum tolerated dose, and recommended dose of the proposed doses of oxaliplatin in this study
* Phase II: To determine the treatment efficacy according to response rates from phase I.

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

Main criteria are listed hereafter:

Inclusion Criteria:

* ECOG: 0-2
* Histological proved rectal adenocarcinoma
* No chemotherapy treatment on the previous 6 months before inclusion.
* No previous pelvic radiotherapy treatment

Exclusion Criteria:

* Important Biological abnormality (renal, hepatic and/or hematological)
* Intestinal occlusion or subocclusion
* Peripheral neuropathy
* Pregnant or breast-feeding women. Potential child-bearing women with a positive pregnancy test.
* Participation in other trials on the previous 4 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2002-10; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Phase I : Maximum Tolerated Dose & Recommended Dose | Days 1, 15, 29
Phase II : Response and resectability rate. | 6 cycles in 6 months

CONTACTS AND LOCATIONS:
Overall Officials: José Mª Taboada, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Barcelona, Spain